CLINICAL TRIAL: NCT03946722
Title: Modified Downregulation for Women With Adenomyosis of the Uterus Prior to Frozen-thawed Embryo Transfer.
Acronym: MODA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/0458
Record Dates: First submitted 2019-05-07; First posted 2019-05-13 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Adenomyosis
Keywords: In vitro fertilisation; Assisted conception; Randomised controlled trial; Down-regulation
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomised controlled trial with two parallel arms. Frozen thawed embryo transfer takes approximately 6 weeks in a standard protocol, including a one week period of downregulation. Downregulation will be extended by five weeks in the modified protocol compared to the standard protocol. Participants will be followed up until the pregnancy outcome is determined, maximum 9 months after embryo transfer.
Masking Description: It will not be possible to perform blinding due to the difference in frequency of administration of medication between the two protocols, therefore an open label method will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard downregulation with GnRH analogue (Other): Participants in this arm will be assigned to the routine IVF protocol currently being used in the investigators' IVF unit, as outlined below, with one week of downregulation. Downregulation is the suppression of the ovaries during an IVF cycle in order to perform controlled ovarian stimulation and prevent premature ovulation.
  Start progesterone (Norethisterone 5mg twice daily orally) on day 14 of downregulation cycle and continue for 11 days. Start GnRH analogue (Buserelin 0.5ml subcutaneously once daily) on day 21 of downregulation cycle and reduce to 0.2ml on day 1 of bleed. Baseline scan on day 1 - 5 of bleed and start oestrogen (Progynova 2mg three times daily orally). Serial scanning from day 10 until endometrial thickness more than 8mm. Once endometrial thickness more than 8mm start progesterone (Cyclogest 400mg twice daily vaginally/rectally and Lubion 25mg twice daily subcutaneously) and proceed to embryo transfer on appropriate day for embryo age.
  Interventions: Drug: GnRH analogue downregulation; Other: Participant questionnaire
- Prolonged downregulation with GnRH analogue (Experimental): Participants in this arm will be exposed to an additional five weeks of downregulation using a GnRH analogue. Downregulation is the suppression of the ovaries during an IVF cycle in order to perform controlled ovarian stimulation and prevent premature ovulation.
  Baseline scan on day 1-5 of bleed and administer GnRH analogue (Leuprorelin acetate 3.75 mg subcutaneously single injection). 28 days later administer second dose of GnRH analogue (Leuprorelin acetate 1.875 mg subcutaneously), and 21 days later start oestrogen (Progynova 2 mg three times daily orally). Serial scanning from day 10 of oestrogen until endometrial thickness more than 8mm. Once endometrial thickness more than 8mm start progesterone (Cyclogest 400mg twice daily vaginally/rectally and Lubion 25mg twice daily subcutaneously) and proceed to embryo transfer on appropriate day for embryo age.
  Interventions: Drug: GnRH analogue downregulation; Other: Participant questionnaire

INTERVENTIONS:
Drug: GnRH analogue downregulation — Downregulation is the suppression of the ovaries during an IVF cycle in order to perform controlled ovarian stimulation and prevent premature ovulation.
  Participants will be exposed to one week of downregulation using a GnRH analogue in the standard downregulation arm and 6 weeks of downregulation using a GnRH analogue in the modified downregulation arm.
Other: Participant questionnaire — Participant will be offered the opportunity to complete an adenomyosis symptom assessment questionnaire at the start of their treatment, and again two months after completion of treatment.

SUMMARY:
1 in 7 couples experience difficulty in conceiving. Many will require in vitro fertilization (IVF). IVF involves an initial period of downregulation to suppress the ovaries and prevent premature ovulation. Hormone injections are then used to stimulate a woman's ovaries to produce eggs which are removed by a minor operation. The harvested eggs are mixed with sperm to create embryos in the laboratory. These embryos are replaced in the womb a few days after they are created (fresh embryo transfer). Any remaining embryos are frozen such that they can be thawed and transferred at a later date (frozen thawed embryo transfer, FTET).

The investigators have previously shown that the presence of moderate or severe adenomyosis significantly reduces the chance of clinical pregnancy after embryo transfer. The purpose of this study is to examine whether it is possible to improve the chance of clinical pregnancy in these women by modifying the IVF protocol they undergo for FTET.

The hypothesis is that a prolonged downregulation regimen for women with adenomyosis would reduce the inflammatory reaction in the endometrium of these women and thus improve the chance of implantation after embryo transfer.

Consenting patients will be offered FTET. Those proceeding will be randomized to one of two protocols (A - standard protocol vs. B - prolonged downregulation protocol). Women will also be offered a questionnaire before and after IVF treatment to assess their adenomyosis symptoms .

The primary outcome of the study is clinical pregnancy defined as an intrauterine pregnancy with a visible heart beat older than 6 weeks gestation. Secondary outcomes include livebirth, pregnancy loss (biochemical pregnancy, miscarriage, ectopic pregnancy, stillbirth, termination of pregnancy), gestational age at delivery, birth weight, neonatal mortality, major congenital anomaly, serious medication reaction, number of frozen embryos available for transfer, number of days to achieve optimal endometrial thickness.

DETAILED DESCRIPTION:
Objectives:

The primary objective is to determine whether modified downregulation before embryo transfer improves the chance of clinical pregnancy after embryo transfer in women with moderate/severe adenomyosis of the uterus. A secondary objective is to evaluate the impact of IVF on adenomyosis-related symptom presence, severity and progression.

Type of trial:

A randomised, controlled, multi-site trial in women with moderate/severe adenomyosis of the uterus undergoing frozen-thawed embryo transfer.

Trial design and methods:

This will be a prospective, randomised controlled study of patients undergoing assisted conception.

Prior to assisted conception all patients are referred for a diagnostic scan. The scan is done in a systematic fashion starting from the uterus in longitudinal plane and measurement of the endometrial thickness. The probe is then rotated to the transverse plane and the uterus scanned from the cervix to the fundus with any uterine pathologies noted and measured in 3 orthogonal planes. A 3D ultrasound volume is then be obtained and saved starting with the uterus in longitudinal view making sure to include all uterine tissue in the 3D volume sweep. Any congenital or acquired uterine anomalies are diagnosed according to published diagnostic criteria. Adenomyosis is diagnosed according to the diagnostic criteria outlined by Exacoustos et al and Naftalin et al and graded for severity according to the number of adenomyosis features present (assign a score of 1 for each of: i) asymmetrical myometrial thickening, ii) parallel shadowing, iii) myometrial cysts, iv) disrupted endometrial myometrial junction, v) endometrial striae, vi) endometrial islands, vii) adenomyoma).

The operator then sweeps to the adnexae, starting from the left, identifies and measures the ovaries in 3 orthogonal planes and documents the antral follicle count. Each ovary is examined for the presence of cysts as well as for mobility and tenderness by gentle pressure with the ultrasound probe. Once the ovaries have been assessed the operator examines the pouch of Douglas for the presence of free fluid as well as any evidence of endometriosis such as obliteration and/or endometriotic nodules as previously described by Holland et al. Videosonography for a period of 5 mins will be performed. Once the ultrasound scan is concluded all information is added to the clinical database.

Patients found to have moderate or severe adenomyosis (4 or more features of adenomyosis as defined by Mavrelos et al) on this scan will be approached by a member of the research team. The researcher will describe the project and provide a copy of the patient information leaflet. Patients will then be invited to return to the unit at a designated time for a scan by a member of the research team. On return to the unit the researcher will repeat the scan to confirm eligibility.

After the scan and once eligibility is confirmed patients will be asked to confirm if they want to participate in the trial. If they agree they will be asked to sign a consent form.

Participating patients will then be followed through the process of assisted conception.

Consenting patients will be randomized to one of two protocols (A vs. B) for frozen thawed embryo transfer.

Protocol A (standard) - start Norethisterone on day 14 of downregulation cycle and continue for 11 days. Start Buserelin 0.5ml on day 21 of downregulation cycle and reduce to 0.2ml on day 1 of bleed. Baseline scan on day 1 - 5 of bleed and start Progynova 2mg TDS PO. Serial scanning from day 10 until endometrial thickness more than 8mm. Once endometrial thickness more than 8mm start cyclogest 400mg BD PV/PR and lubion 25mg BD and proceed to embryo transfer on appropriate day for embryo age.

Protocol B (modified) - Baseline scan on day 1-5 of bleed and administer Triptorelin acetate 3.75 mg. 28 days later administer 1.875 mg Triptorelin acetate and 21 days later start Progynova 2 mg TDS PO. Serial scanning from day 10 of Progynova until endometrial thickness more than 8mm. Once endometrial thickness more than 8mm start Cyclogest 400mg BD PV/PR and Lubion 25mg BD and proceed to embryo transfer on appropriate day for embryo age.

Patients will be offered the opportunity to complete an adenomyosis symptom assessment questionnaire at the start of their treatment, and again two months after completion of treatment.

Trial duration per participant:

8-12 weeks

Estimated total duration:

3 years.

Planned trial sites:

Multi-site.

Total number of participants planned:

162.

Sample size estimation:

The investigators recently reported that the clinical pregnancy rate in women with moderate to severe adenomyosis is 22.9% vs. 42.7% in women with mild disease. They speculate that the modified protocol will improve the chance of clinical pregnancy to be equivalent to those with mild disease.

162 patients are required to have an 80% chance of detecting an increase in the clinical pregnancy rate from 22.9% in the control group to 42.7% in the experimental group, as significant at the 5% level (α = 0.05, β = 0.20). The trial is powered at 80%.

Statistical methodology and analysis:

The investigators will first perform univariate analysis to explore significant differences in the demographic characteristics (age, duration of subfertility), and clinical factors known to impact the outcome of assisted conception (number of oocytes retrieved, number and quality of embryos transferred) between women randomized to standard and modified FTET protocol.

In the second stage analysis the investigators will perform univariate analysis to compare the primary outcome (clinical pregnancy rate after FTET) between woman randomized to the standard and modified clinical protocol. The investigators will perform univariate analysis to compare secondary outcomes (livebirth, pregnancy loss (biochemical pregnancy, miscarriage, ectopic pregnancy, stillbirth, termination of pregnancy), gestational age at delivery, birth weight, neonatal mortality, major congenital anomaly, serious medication reaction, number of frozen embryos available for transfer, number of days to achieve optimal endometrial thickness). They will perform a sub-analysis for women with co-existing endometriosis. All models will be estimated in the Stat 12 statistical software.

ELIGIBILITY:
Inclusion Criteria:

1. Couples who are undergoing a cycle of IVF/ICSI, where a cycle is defined as egg collection following ovarian stimulation.
2. The female partner is ≥18 and < 42 years of age.
3. The female partner has a BMI <30.
4. Two out of three of the following criteria are met: AMH >5.4, FSH <8.9, antral follicle count >4.
5. Moderate or severe adenomyosis of the uterus diagnosed on ultrasound scan.
6. Both partners are willing and able to provide written informed consent.

Exclusion Criteria:

1. Concurrent and/or recent involvement in other research that is likely to interfere with the intervention within the previous 3 months of study enrolment.
2. Previous open or laparoscopic myomectomy
3. Uterine fibroids (untreated FIGO Type 0-I-II and type III-IV fibroids > 3 cm)
4. Use of GnRH analogues within previous 3 months.
5. Severe male factor infertility (sperm count < 2 x 106/ml, use of surgically retrieved spermatozoa)
6. Couples who in the opinion of the researcher by virtue of language or learning impairment would be unable to give fully informed consent to the study.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Adenomyosis of the uterus is a condition which affects women only.
Enrollment: 162 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2023-08-17 (Estimated); Study Completion 2024-05-17 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 weeks after embryo transfer
  Clinical pregnancy is defined as an intrauterine pregnancy with a visible heart beat older than 6 weeks gestation.

SECONDARY OUTCOMES:
Livebirth | 9 months after embryo transfer
  Pregnancy greater than 24 weeks
Pregnancy loss | 9 months after embryo transfer
  Includes biochemical pregnancy, miscarriage, ectopic pregnancy, stillbirth, termination of pregnancy
Gestational age at delivery | 9 months after embryo transfer
  Number of weeks at which infant is delivered
Birthweight at delivery | 9 months after embryo transfer
  Weight at time of delivery
Neonatal mortality | 9 months after embryo transfer
  The death of a baby before or during birth after 24 weeks of gestation
Major cogenital anomaly | 9 months after embryos transfer
  Major cogenital anomaly
Serious medication reaction | 9 months after embryo transfer
  Serious medication reaction
Number of frozen embryos available for transfer | Day of embryo transfer
  Number of frozen embryos available for transfer
Number of days to achieve optimal endometrial thickness | Start of endometrial preparation until day of embryo transfer
  Number of days to achieve optimal endometrial thickness
Presence and severity of adenmyosis-related symptoms | 2 months after embryo transfer
  Menorrhagia, dysmenorrhoea

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of the research group.

REFERENCES:
- [Derived] Latif S, Wattar BHA, Balachandren N, Lukaszewski T, Saridogan E, Yasmin E, Serhal P, Mavrelos D. Effectiveness of modified downregulation for women with moderate and severe adenomyosis of the uterus prior to frozen thawed embryo transfer (MODA) study protocol: a pragmatic randomised-controlled trial. BMJ Open. 2021 Oct 29;11(10):e050248. doi: 10.1136/bmjopen-2021-050248. PMID 34716161